CLINICAL TRIAL: NCT04021719
Title: OnTrackNY's Learning Healthcare System
Status: Suspended | Type: Observational
Why Stopped: U.S. Department of Health and Human Services OHRP issued an FWA restriction on NYSPI research that included a pause of human subjects research as of June 23, 2023. This study will resume recruitment after OHRP has approved the resumption of research.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other); New York University (Other); Washington University School of Medicine (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lisa Dixon, Clinical Professor, New York State Psychiatric Institute
Other Study IDs: 7840; 5R01MH120597 (NIH)
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: First Episode Psychosis
Keywords: First Episode Psychosis; Learning Healthcare system; Stakeholders; Data infrastructure; Psychotic disorders; Mental disorders; Schizophrenia Spectrum and Other Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders; Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OnTrackNY LHS Participants and Stakeholders: OnTrackNY participants and stakeholders, including past participants, family members, clinicians, administrators, payors, and state leadership
  Interventions: Other: Stakeholder feedback; Other: Data infrastructure

INTERVENTIONS:
Other: Stakeholder feedback — Stakeholders, including OnTrackNY participants, past participants, family members, clinicians, administrators, payors and state leadership, will participate in a variety of activities to provide continuous quality improvement to the OnTrackNY program, including a Stakeholder Workgroup, interviews and focus groups
Other: Data infrastructure — Data will be systematically collected as part of CQI activities, within a state-of-the-art data infrastructure that allows for client-level feedback to clients, providers and sites to improve quality of care.

SUMMARY:
This application proposes OnTrackNY as a regional scientific hub for the Early Psychosis Intervention Network (EPINET) program as part of the National Institute of Mental Health (NIMH)'s creation of a national learning health care system (LHS) for early psychosis care. OnTrackNY has grown into a 22-site network, under the leadership of Lisa Dixon, MD, MPH.

Created and supported by the New York State's Office of Mental Health (OMH), OnTrackNY is a nationally recognized model providing coordinated specialty care (CSC) for adolescents and young adults within two years of the onset of non-affective psychosis. OMH regulates and licenses all mental health programs in New York and is a direct-services provider via state-operated programs statewide. This makes OMH an ideal partner for establishing a statewide learning health care system for early psychosis care. Further, OnTrackNY's administration, OnTrackCentral, operates within the OMH-supported Center for Practice Innovations at Columbia Psychiatry. In this model, OnTrackCentral serves as the hub and the 22 OnTrackNY programs serve as the spokes. Since 2014, the still-growing OnTrackNY network has served over 1,600 individuals. From its inception, OnTrackNY has aimed to deliver high-quality, data-driven, accountable and culturally competent care consistent with an LHS. As a condition of funding, all OnTrackNY providers follow established protocols that require submission of patient- and site-level standard measures of early psychosis clinical features, services, and treatment outcomes.

The proposed EPINET regional hub, the OnTrackNY LHS, will emphasize and enhance two critical foundational components - Aim 1: proactively engage stakeholders to optimize understanding of key problems and their solutions at every LHS phase; and Aim 2: develop data systems with enhanced standardized data collection, including post-discharge data and linkages to external data systems, and enhancing data analytics that will allow for client-level treatment planning and prospective analytics, delivering real time, dynamic and actionable information to stakeholders. These LHS components do not follow in a stepwise sequence but instead operate in parallel and interact to facilitate and enhance quality improvement processes. This backbone will support the development of practice-based research.

DETAILED DESCRIPTION:
This application proposes OnTrackNY as a regional scientific hub for the Early Psychosis Intervention Network (EPINET) program as part of NIMH's creation of a national learning health care system (LHS) for early psychosis care. As a continuation of the NIMH-supported RAISE-Implementation and Evaluation Study, OnTrackNY has grown into the 22-site (and still expanding) network under the leadership of Lisa Dixon, MD, MPH. OnTrackNY is a nationally recognized model for providing CSC for adolescents and young adults within two years of the onset of non-affective psychosis. OnTrackNY sites are located in licensed outpatient clinics at community agencies, state-operated facilities, and community and academic hospitals in urban, suburban, and rural areas throughout New York. This network has served over 1,600 individuals to date, with 451 new enrollees in calendar year 2017. Thanks to its sponsorship by the New York State Office of Mental Health (OMH), OnTrackNY has progressed to meet its goal of providing CSC to any young person with early psychosis in New York State, regardless of ability to pay. OnTrackNY includes OnTrackCentral-the "hub"-a team of nine staff, who provide training and technical assistance to sites and manage data collection, and the 22 teams which are its "spokes." From its inception, OnTrackNY has sought to deliver high-quality, data-driven, accountable care consistent with an LHS. (See Facilities for details on sites.)

The Foundations of a LHS in OnTrackNY: Several factors facilitated OnTrackNY's LHS foundations: 1) OnTrackNY evolved from the data-oriented RAISE-Implementation and Evaluation Study; 2) its location within the Center for Practice Innovations, an OMH-funded and empirically driven technical assistance center for scaling up evidence-based practices housed within Columbia Psychiatry; and 3) a strong commitment by OMH to high quality, accountable care. OnTrackCentral obtains stakeholder input from clinicians, program directors and state administrators. All OnTrackNY teams are contractually obligated to follow established protocols requiring specific service components and standardized client- and site-level measures for treating first episode psychosis (FEP). OnTrackCentral provides ongoing technical assistance to support the model, identify programmatic gaps and problems, and facilitate practice-based learning and research.

The Opportunity for OnTrackNY to Build a Better LHS: EPINET provides the opportunity to leverage the nascent LHS foundations of OnTrackNY and build a large, state-of-the-art LHS for early psychosis care. The investigators propose to expand and restructure the continuous quality improvement (CQI) process to: (Aim 1) include key stakeholders at every phase of the LHS and (Aim 2) provide accurate and appropriate delivery of real-time data to clients and providers to facilitate measurement-based care.

LHS Frameworks and Conceptual Model: This LHS is based on the principles of the Institute of Medicine's (IOM) (now National Academy of Medicine) model for a continuously learning healthcare system which brings together stakeholders to review data and technologies to develop and apply strategies to improve quality and increase efficiency. The investigators will use the IOM's LHS model, operationalizing the components according to the six LHS phases described by the Group Health Cooperative. While this LHS model provides an aspirational roadmap for a cyclic improvement approach, significant knowledge gaps limit translation and implementation of knowledge into evidence-based communications, campaigns, guidelines and other tools, products, and interventions. The investigators will draw on the Knowledge to Action (KTA) framework, which guides knowledge translation and implementation activities within each phase of the LHS model. The KTA planning tool directs knowledge creation and action cycles through questions for stakeholders to consider during each LHS phase. Through an iterative process, knowledge creation begins with stakeholders, data and mixed methods practice- based research during the LHS Scanning and Surveillance phase. The Action Cycle outlines a process, representing the activities needed for knowledge to be implemented in practice. Knowledge is adapted to the local context, and barriers and facilitators to its use are explicitly assessed. Stakeholders are centrally involved in tailoring knowledge and interventions to those who will use it.

This proposal will thus build a stakeholder-driven LHS that will establish the data infrastructure needed to promote measurement-based treatment within a structure supporting continuous quality improvement which, in turn, supports practice-based research-with the overall goal of improving care and outcomes for individuals with early psychosis. This EPINET-supported LHS will create an engine to optimize the potential of CSC to improve the lives of people with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* OnTrackNY participants are individuals age 16-30 who have experienced non-affective psychoses for less than two years and have enrolled at an OnTrackNY site. Other stakeholders include past OnTrackNY participants, family members, clinicians, administrators, payors and agency leadership.

Exclusion Criteria:

* Not meeting inclusion criteria specified above

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: OnTrackNY participants at an OnTrackNY site (currently 28 sites statewide) or other stakeholders.
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Participation in work and school | Up to 5 years
  Participation in competitive employment and/or degree-based education program, as assessed in OnTrackNY assessment instruments
MIRECC GAF occupational, social and symptom functioning | Up to 5 years
  Improvements in occupational, symptom and social functioning, as measured by the MIRECC Global Assessment of Functioning (GAF) scores
Hospitalization rates | Up to 5 years
  Decreases in rates of psychiatric hospitalization per quarter, as assessed in OnTrackNY assessment instruments

CONTACTS AND LOCATIONS:
Overall Officials: Lisa B Dixon, MD, MPH, Principal Investigator — New York State Psychiatric Institute; Iruma Bello, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- OnTrackNY Central, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel SR, Bello I, Cabassa LJ, Nossel IR, Wall MM, Montague E, Rahim R, Mathai CM, Dixon LB. Adapting coordinated specialty care in the post-COVID-19 era: study protocol for an integrative mixed-methods study. Implement Sci Commun. 2021 Jul 5;2(1):72. doi: 10.1186/s43058-021-00178-x. PMID 34225817
- [Derived] Patel S, Bello I, Cabassa LJ, Nossel IR, Wall MM, Montague E, Rahim R, Mathai CM, Dixon LB. Adapting Coordinated Specialty Care in the Post-COVID-19 Era: Study Protocol for an Integrative Mixed-methods Study. Res Sq [Preprint]. 2021 Apr 26:rs.3.rs-452200. doi: 10.21203/rs.3.rs-452200/v1. PMID 34013257